CLINICAL TRIAL: NCT00511420
Title: Effects of Cocoa Products on Cardiovascular Disease Risk Factors
Acronym: CoCD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Cocoa products; Ministerio de Educacion
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular Diseases
Keywords: cocoa; cardiovascular disease; blood pressure
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Cocoa and other ingredients (product type 1). This product is a control of type 2.
  Interventions: Dietary Supplement: Cocoa product type 1
- 2 (Placebo Comparator): Cocoa plus hazelnuts and other ingredients (product type 2). This product is a control of type 3 and 4.
  Interventions: Dietary Supplement: Cocoa product type 2
- 3 (Active Comparator): Cocoa plus hazelnuts and other ingredients (cocoa product type 3).
  Interventions: Dietary Supplement: Cocoa product type 3
- 4 (Active Comparator): Cocoa, hazelnuts and other ingredients called LMN (cocoa product type 4).
  Interventions: Dietary Supplement: Cocoa product type 4

INTERVENTIONS:
Dietary Supplement: Cocoa product type 1 — 6 doses of 13 grams per day during 4 weeks with a prior stabilization period of 2 weeks.
  Arms: 1
Dietary Supplement: Cocoa product type 2 — 6 doses of 13 grams per day during 4 weeks with a prior stabilization period of 2 weeks with cocoa product type 1
  Arms: 2
Dietary Supplement: Cocoa product type 3 — 6 doses of 13 grams per day during 4 weeks with a prior stabilization period of 2 weeks with cocoa product type 1
  Arms: 3
Dietary Supplement: Cocoa product type 4 — 6 doses of 13 grams per day during 4 weeks with a prior stabilization period of 2 weeks with cocoa product type 1
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the effects of optimized composition chocolates that include natural ingredients with demonstrated biological activity are observed cardioprotectores effects in the human.

DETAILED DESCRIPTION:
Studies carried out during the last decades have demonstrated of conclusive form that foods like nuts, products like cocoa or other ingredients, to be consumed of isolated form or when taking several from integrated them in a same diet can contribute to the prevention or the treatment of the cardiovascular diseases.

The study was a randomized, controlled, double-blind, parallel multi-center study in which the 4 different types of cocoa products [1)cocoa and other ingredients (sugar and vegetal oils), 2)cocoa plus hazelnuts and other ingredients, 3)the same as 2 plus other ingredient and 4) cocoa, hazelnuts and other ingredients called (LMN)], introduced into a calorie-balanced diet for 4 weeks with a prior stabilization period of 2 weeks in which all participants received the cocoa product type 1. Cocoa product type 1 is a control of type 2, and types 1 and 2 were controls of types 3 and 4.

Cocoa products type 4 is registered as patent. The trial was conducted in Reus and 3 other cities in Catalonia (Alcover, Centelles and Vic) (Spain).

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants had systolic blood pressure (BP) of 120 to 159 mm Hg or a diastolic blood pressure of 80 to 99 mm Hg. This range includes participants with prehypertension (systolic, 120-139 mm Hg or diastolic, 80-89 mm Hg) and stage 1 hypertension (systolic, 140-159 mm Hg or diastolic, 90-99 mm Hg).
* Moreover, participants' plasma LDL-cholesterol concentrations were ≥ 3.35 mmol/L (≥ 130 and ≤ 189 mg/dL) and triglyceride concentrations < 4 mmol/L (350 mg/dL) in the fasting state and at least one CVD risk factor such as age (men ≥45 years; women ≥55 years), cigarette smoking, low high density lipoprotein cholesterol concentration (<1.0 mmol/L (40 mg/dL) and <1,18 mmol/L (46 mg/dL), men and women, respectively), family history of premature CVD (in male first-degree relative <55 years of age, in female first-degree relative <65 years of age.

Exclusion Criteria:

* Assessed from the medical history and a complete physical examination, were plasma triglyceride concentrations ≥4 mmol/L (350 mg/dL), BMI >35 kg/m2, CVD clinical events, use of lipid-lowering drugs at least 2 months prior to the start of study, diabetes mellitus (at least 2 fasting glucose ≥7.0 mmol/L (≥ 126 mg/dL), renal insufficiency, thyroid or other endocrine disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2005-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure changes between baseline and the end of intervention | 4 weeks

SECONDARY OUTCOMES:
Plasma lipids, lipoproteins and apolipoproteins | 4 weeks
Endothelial dysfunction, oxidation and inflammation markers | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Sola, Dra/Prof, Principal Investigator — University Rovira i Virgili; Bartolome Ramirez, Mr, Principal Investigator — La Morella Nuts, S.A.
Locations (1):
- Universitat Rovira i Virgili and Hospital Universitari Sant Joan, Reus, Tarragona, Spain

REFERENCES:
- [Derived] Crescenti A, Sola R, Valls RM, Caimari A, Del Bas JM, Anguera A, Angles N, Arola L. Cocoa Consumption Alters the Global DNA Methylation of Peripheral Leukocytes in Humans with Cardiovascular Disease Risk Factors: A Randomized Controlled Trial. PLoS One. 2013 Jun 26;8(6):e65744. doi: 10.1371/journal.pone.0065744. Print 2013. PMID 23840361
- [Derived] Sola R, Valls RM, Godas G, Perez-Busquets G, Ribalta J, Girona J, Heras M, Cabre A, Castro A, Domenech G, Torres F, Masana L, Angles N, Reguant J, Ramirez B, Barriach JM. Cocoa, hazelnuts, sterols and soluble fiber cream reduces lipids and inflammation biomarkers in hypertensive patients: a randomized controlled trial. PLoS One. 2012;7(2):e31103. doi: 10.1371/journal.pone.0031103. Epub 2012 Feb 27. PMID 22383996